CLINICAL TRIAL: NCT06804772
Title: A Clinical Study to Evaluate the Efficacy of Activated Silk™ 27P-α to Improve the Signs of Aging, Part 2
Brief Title: A Clinical Study to Evaluate the Efficacy of Activated Silk™ 27P-α in Subjects, Aged 35-65 Years of Age, to Improve the Signs of Aging, by Comparing to a Placebo
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Victoria Collotta (Industry)
Responsible Party: Sponsor-Investigator, Victoria Collotta, General Manager, Branded Products, Principal Investigator, Evolved By Nature
Organization: Evolved By Nature (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: Single | Purpose: Other
Other Study IDs: CLN-SKN02-011
Record Dates: First submitted 2025-01-16; First posted 2025-02-03 (Actual); Last update posted 2025-02-03 (Actual); Status verified 2024-12

CONDITIONS: Skin Aging

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- ~15 subjects, aged 35-65, will receive Investigational Facial Serum #3 (Placebo Comparator)
  Interventions: Other: Investigational Facial Serum #3
- 0 female subjects, aged 35-65, will receive Investigational Facial Serum #1 (Experimental)
  Interventions: Other: Investigational Facial Serum #1
- 0 female subjects, aged 35-65 years of age, will receive Investigation Facial Serum #2 (Active Comparator)
  Interventions: Other: Investigational Facial Serum #2

INTERVENTIONS:
Other: Investigational Facial Serum #3 — Investigational Facial Serum #3 is a placebo comparator
  Arms: ~15 subjects, aged 35-65, will receive Investigational Facial Serum #3
Other: Investigational Facial Serum #1 — Investigational Facial Serum #1 is made with Activated Silk™ 27P-α.
  Arms: 0 female subjects, aged 35-65, will receive Investigational Facial Serum #1
Other: Investigational Facial Serum #2 — Investigational Facial Serum #2 is made with an active comparator.
  Arms: 0 female subjects, aged 35-65 years of age, will receive Investigation Facial Serum #2

SUMMARY:
A clinical study with approximately 15 subjects, aged 35-65 years of age, who must have crow's feet and at least one other type of facial fine lines/wrinkles in order to evaluate the efficacy of Activated Silk™ 27P-α to improve the signs of aging, by comparing to a placebo.

ELIGIBILITY:
Inclusion Criteria:

* Healthy individuals, between the ages of 35 - 65 years of age, with no known medical conditions that interfere with study participation, are the priority.
* Subject has signed a written Informed Consent prior to Day -7.
* 100% of subjects have crow's feet and at least one of the following: forehead lines/wrinkles (e.g. vertical lines between eyebrows, horizontal lines above the eyebrow), marionette lines, nasolabial folds.
* 50% of subjects have self-perceived sensitive skin.
* 20% of the subjects are not 100% Caucasian.

Exclusion Criteria:

* Subject is pregnant, nursing, or planning to become pregnant.
* Subject is currently using medication likely to affect the response to investigational formulation.
* Subject had a fever in the last 12 hours prior to the start of the study.
* Subject has a pacemaker or significant medical history of hepatic, renal, cardiac, pulmonary, digestive, hematological, neurological, locomotor or psychiatric disease; cancer; multiple sclerosis; high blood pressure; thrombosis; phlebitis; insulin-dependent diabetes; or any such related medical condition(s) that may interfere with the completion of the study.
* The Subject used a form of retinol on their face in the past six months.
* The Subject used any prescription skincare products on their face in the last six months.
* The Subject has received any laser, chemical peel, or other facial resurfacing treatment such as microdermabrasion, dermablading or microneedling in the past four weeks.
* The Subject received Botox, Dysport, other muscle relaxers or injectable skin fillers in the face during the past six months.
* Subject has a known allergy or sensitivity to any ingredient in the aqueous skincare formulation provided for their use in the trial .
* Subject is currently participating in another study utilizing facial products.
* Subject is blind, visually impaired or decisionally impaired.

Ages: 35 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2024-12-03 (Actual); Primary Completion 2025-01-03 (Actual); Study Completion 2025-01-31 (Estimated)

PRIMARY OUTCOMES:
Change in appearance of fine lines/wrinkles as evaluated by the Principal Investigator using a scale from 0-9 | Day 0 to Day 28
  Change in appearance of fine lines/wrinkles for subjects treated with Investigational Facial Serum #3 at Day 28 vs. Day 0

SECONDARY OUTCOMES:
Change in appearance of skin characteristics | Day 0 to Day 28
  Change in surface hydration as measured by the Corneometer for subjects treated with Investigational Facial Serum #3 at Day 14 and Day 28 vs. Day 0
Change in appearance of skin characteristics | Day 0 to Day 28
  Change in transepidermal water loss as measured by the Tewometer for subjects treated with Investigational Facial Serum #3 at Day 14 and Day 28 vs. Day 0.

CONTACTS AND LOCATIONS:
Locations (1):
- Evolved By Nature, Needham, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No